CLINICAL TRIAL: NCT02621957
Title: A Phase 1, Open-Label Study to Evaluate the Effect of GDC-0810 on the Pharmacokinetics of Pravastatin in Healthy Female Subjects of Non-Childbearing Potential
Brief Title: Effect of GDC-0810 on the Pharmacokinetics of Pravastatin in Healthy Female Subjects of Non-Childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GP29825
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 3-(4-(2-(2-chloro-4-fluorophenyl)-1-(1H-indazol-5-yl)but-1-en-1-yl)phenyl)acrylic acid; Pravastatin

ARMS (1):
- Female Healthy Volunteers (Experimental): Healthy volunteer female subjects of non-childbearing potential will be administered pravastatin once on Day 1 during Period 1 (Day -1 to Day 4). During Period 2 (Days 5-28) GDC-0810 will be administered daily on Days 5-8. Pravastatin will be co-administered on Day 7.
  Interventions: Drug: GDC-0810; Drug: Pravastatin

INTERVENTIONS:
Drug: GDC-0810 — During Period 2 subjects will be administered an oral 600 mg dose GDC-0810 daily beginning on Day 5 for 4 consecutive days (from Days 5 to 8, inclusive).
  Other Names: ARN-810
Drug: Pravastatin — Subjects will receive a single oral dose of 10 mg pravastatin on Day 1 in Period 1 and Day 7 in Period 2.
  Other Names: Pravachol

SUMMARY:
This study is to assess the pharmacokinetics (PK) of a single dose of pravastatin with and without concomitant GDC-0810 administration in healthy female subjects of non-childbearing potential. During Period 1 (Day -1 to Day 4) PK parameters of pravastatin will be determined in the absence of GDC-0810. During Period 2 (Days 5-28) PK parameters of pravastatin will be determined in the presence of GDC-0810.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between 18 and 65 years of age, inclusive.
* Female subjects of non-childbearing potential including non-pregnant, non-lactating, and either postmenopausal or surgically sterile for at least 45 days post procedure.
* Within BMI range 18.5 to </= 29.9 kg/m^2, inclusive.
* In good health, as determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory evaluations.
* Receive an explanation of the mandatory pharmacogenomic (PgX) component of the study.

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder.
* Previous history of adverse reaction to statins.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days or 5 half-lives, whichever is longer, prior to Check-in (Day -1) in Period 1.
* Use of systemic hormone replacement therapy within 1 year prior to Check-in (Day -1).
* History of use of tamoxifen, aromatase inhibitor or any other endocrine agent for treatment of breast cancer.
* Female subject is pregnant lactating, or breast feeding.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Time to Maximum Concentration (Tmax) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Area Under the Concentration-Time Curve from Hour 0 to the Last Measurable Concentration (AUC0-t) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Area Under the Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Apparent Volume of Distribution (Vz/F) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Apparent Clearance (CL/F) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Apparent Terminal Elimination Rate Constant (lambda z) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Apparent Terminal Elimination Half-Life (t1/2) of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)
Amount of Pravastatin Excreted in Urine (Ae) | Day 1 (Period 1) and Day 7 (Period 2)
Renal Clearance (CLR) of Pravastatin | Day 1 (Period 1) and Day 7 (Period 2)
Percentage of Pravastatin Excreted in Urine (%Excreted) | Day 1 (Period 1) and Day 7 (Period 2)
Plasma Concentrations of Pravastatin | Days 1-3 (Period 1) and Days 7-10 (Period 2)

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of GDC-0810 | Days 7-10 (Period 2)
Time to Maximum Concentration (Tmax) of GDC-0810 | Days 7-10 (Period 2)
Area Under the Concentration-Time Curve from Hour 0 to the Last Measurable Concentration (AUC0-t) of GDC-0810 | Days 7-10 (Period 2)
Area Under the Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of GDC-0810 | Days 7-10 (Period 2)
Apparent Volume of Distribution (Vz/F) of GDC-0810 | Days 7-10 (Period 2)
Apparent Clearance (CL/F) of GDC-0810 | Days 7-10 (Period 2)
Apparent Terminal Elimination Rate Constant (lambda z) of GDC-0810 | Days 7-10 (Period 2)
Apparent Terminal Elimination Half-Life (t1/2) of GDC-0810 | Days 7-10 (Period 2)
Amount of GDC-0810 Excreted in Urine (Ae) | Day 7 (Period 2)
Renal Clearance (CLr) of GDC-0810 | Day 7 (Period 2)
Percentage of GDC-0810 Excreted in Urine (%Excreted) | Day 7 (Period 2)
Percentage of Participants with Adverse Events (AEs) | From baseline to study completion up to Day 28
Percentage of Participants with Serious Adverse Events (SAEs) | From baseline to study completion up to Day 28
Percentage of Participants with Clinically Significant Changes in Safety Measurements, Including Vital Signs, Electrocardiograms (ECGs), Physical Examination Findings and Clinical Laboratory Results. | From baseline to study completion up to Day 28
Plasma Concentrations of GDC-0810 | Days 7-10 (Period 2)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Daytona Beach, Florida, United States